CLINICAL TRIAL: NCT04081129
Title: Using EIT to Assess the Effect of Early Mobilization on Regional Lung Ventilation in ICU Patients
Brief Title: Effect of Early Mobilization on Regional Lung Ventilation Assessed by EIT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Yun Long (Other)
Responsible Party: Sponsor-Investigator, Yun Long, the director of the intensive care medicine, Peking Union Medical College Hospital
Organization: Peking Union Medical College Hospital (Other)
Other Study IDs: EIT-early mobilization
Record Dates: First submitted 2019-09-03; First posted 2019-09-09 (Actual); Last update posted 2019-09-10 (Actual); Status verified 2019-09

CONDITIONS: Critical Illness; Lung Function Decreased; ICU Acquired Weakness
Keywords: EIT; early mobilization
MeSH Terms: conditions — Critical Illness; Respiratory Insufficiency

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- ICU patients with early mobilization

SUMMARY:
Changes in pulmonary ventilation and perfusion by EIT to out-of-bed activity in critically ill patients

DETAILED DESCRIPTION:
1. EIT measurements were performed in ICU patients who under out-of-bed activity
2. Measurement of EIT was taken place at 4 time points: supine position before early mobilization, 30min, 60min during early mobilization, supine positon after early mobilization. All of them were without invasive ventilation. Measurements were made in triplicate at all time points.

ELIGIBILITY:
Inclusion Criteria:

* adult patients was performed out-of-bed activity in the ICU department based on doctor order
* Age (> 18 years old) and (< 90 years old)

Exclusion Criteria:

* Chest skin is injury and cannot be monitored by EIT
* The patients or their families refused to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: adult patients was performed out-of-bed activity, who were sequentially admitted to the ICU
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2019-12-31 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
lung regional ventilation distribution | Hour 1
  lung regional ventilation distribution was measured by EIT

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Yuan S, Chi Y, Long Y, He H, Zhao Z. Effect of Position Change From the Bed to a Wheelchair on the Regional Ventilation Distribution Assessed by Electrical Impedance Tomography in Patients With Respiratory Failure. Front Med (Lausanne). 2021 Nov 4;8:744958. doi: 10.3389/fmed.2021.744958. eCollection 2021. PMID 34805212